CLINICAL TRIAL: NCT06404008
Title: A Controlled Breathing Intervention to Reduce Stress and Improve Symptoms in COPD Patients (REST): A Randomized Pilot Trial
Brief Title: A Controlled Breathing Intervention to Reduce Stress and Improve Symptoms in COPD Patients (REST)
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Trisha M. Parekh, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005553
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: COPD; Stress; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Educational Status

STUDY DESIGN:
Masking Description: Only the statistician will be blinded to study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (REST) (Experimental): Participants randomized to this group will receive COPD education, research staff support, and the REST (controlled breath) intervention.
  Interventions: Behavioral: REST
- Control (Active Comparator): Participants randomized to this group will receive COPD education and research staff support.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: REST — After randomization, individuals will attend an in-person training session in the REST protocol. This is a 15 minute controlled breath protocol that includes 3 yoga breathing techniques: 3-part dirgha breath, alternate nostril breathing, and 2:1 breathing. Each technique will be completed for 5 minutes, for a total of 15 minutes. After the training session, participants will practice the REST protocol for 15 minutes twice a day with guidance from research staff over zoom (Days 1-7) with daily COPD education including inhaler technique, nutrition, vaccinations, tobacco cessation counseling, and exacerbation education. On Day 8, participants will attend the Trial Session where they will complete the REST protocol (15 minutes) while vitals, lung function, and ECG measurements are taken. Surveys will be administered before and after the REST protocol to document patient reported stress and dyspnea.
  Arms: Behavioral Intervention (REST)
Other: Education — After randomization, individuals will attend an in-person education session led by a research coordinator. For the following 7 days, the research staff will call patients daily and provide daily COPD education including inhaler technique, nutrition, vaccinations, tobacco cessation counseling, and COPD exacerbation education. On Day 8, participants will attend the Trial Session where they will do spontaneous breathing (15 minutes) while vitals, lung function, and EKG measurements are taken. Surveys will be administered before and after the spontaneous breathing period to document patient reported stress and dyspnea. After the study, participants will be asked to complete a close out survey and interview over zoom.
  Arms: Control

SUMMARY:
This is a parallel design, randomized, controlled pilot trial comparing a controlled breath intervention (REST) to usual care for reducing stress in individuals with COPD.

DETAILED DESCRIPTION:
This is a parallel design, randomized, controlled pilot trial comparing a controlled breath intervention (REST) to usual care for reducing stress in individuals with chronic obstructive pulmonary disease (COPD). The intervention is based on the breathing techniques of Pranayama. It was developed with patient and stakeholder input and is targeted for individuals with COPD who have moderate levels of stress and symptom burden. The intervention is a 15-minute breathing protocol which will be taught to participants and subsequently evaluated in a clinic setting with surveys, lung function, and cardiac assessments. This intervention will be pre-tested in 6 individuals, revised, and piloted in 30 individuals (15 in intervention group, 15 in control group). This study will answer the question of 1) whether a controlled breath protocol is feasible, acceptable, and safe for patients with COPD and 2) whether any modifications to the intervention are needed for a future multicenter trial to be proposed and conducted after the completion of the pilot trial. We will also 3) obtain sufficient estimates of variability in stress measures to inform statistical planning of a future trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spirometry confirmed COPD (FEV1/FVC <0.70 + FEV1<80%)
* Perceived Stress Scale > 13
* Age >40 years old
* Able to read, write, and speak in English
* Able to attend 1 in person training session and 1 in person trial sessions

Exclusion Criteria:

* Current regular practice of breathing exercises or pranayama
* No access to internet or telephone
* Recent hospitalization for COPD exacerbation or any reason in the past 30 days
* Other primary lung disease (ILD, asthma, bronchiectasis) by self-report or chart review
* Non-correctable hearing impairment (i.e. hearing impairment despite hearing aids)
* Severe cognitive impairment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility | 6 months
  IG: Completion of 2 in-person sessions (1 training, 1 trial) along with >80% of daily individual practice of breathing protocol (15 minute twice daily)
Trial feasibility | 6 months
  Rates of screening, enrollment, retention, reasons for exclusion and refusals, and attrition. Attrition goal <10% throughout study period.
Acceptability (quantitative) | 6 months
  Post-intervention survey on intervention acceptability with Likert scale rated 1 to 10; 10 being most acceptable. Overall average score ≥8 of 10 defined as acceptable. Will assess patient reported enjoyment, difficulty, and adherence
Acceptability (qualitative) | 6 months
  Post-intervention semi-structured, in-depth interviews by telephone conducted by study coordinator to explore acceptability, barriers, facilitators, and survey burden

SECONDARY OUTCOMES:
Perceived Stress Scale | Day 0, Day 8
  10-item questionnaire with a score of 0-40, with higher scores indicating higher levels of stress.
Modified Medical Research Council dyspnea scale | Day 0, Day 8
  Self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4
Mindful Attention Awareness Scale | Day 0, Day 8
  The MAAS is a 15-item scale designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present

OTHER OUTCOMES:
Lung Function | Day 0, Day 8
  Forced expiratory volume in 1 second (L), Forced vital capacity, Inspiratory capacity
Heart rate variability | Day 0, Day 8
  Derived from 10-second ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Ascension Seton Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No